CLINICAL TRIAL: NCT03227445
Title: A Randomized, Open-label, Cross-over, Placebo Inhaler Study to Evaluate the Correct Use of ELLIPTA™ Dry Powder Inhaler (DPI) Compared to DISKUS™ DPI Used in Combination With HandiHaler DPI in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Comparative Study of ELLIPTA Dry Powder Inhaler (DPI) Versus DISKUS DPI Used With HandiHaler DPI in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206901
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: DISKUS; HandiHaler; COPD; Placebo; Cross-over; Dry powder inhaler; ELLIPTA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive a placebo ELLIPTA inhaler QD or a placebo DISKUS BID with placebo HandiHaler QD inhaler at Visit 1 and Visit 2 in a cross-over manner followed by Preference Questionnaire 1 or 2
Masking Description: This will an open-label study and blinding will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Treatment sequence A (Experimental): Eligible subjects will use ELLIPTA DPI QD for 28 days in Period 1 followed by DISKUS BID with HandiHaler QD use for 28 days in Period 2. These subjects will then be asked to complete preference questionnaire 1 at Visit 3 (Day 56).
  Interventions: Device: ELLIPTA placebo DPI; Device: DISKUS placebo DPI; Device: HandiHaler placebo DPI; Other: Inhaler preference questionnaires
- Treatment sequence B (Experimental): Eligible subjects will use ELLIPTA DPI QD for 28 days in Period 1 followed by DISKUS BID with HandiHaler QD use for 28 days in Period 2. These subjects will then be asked to complete preference questionnaire 2 at Visit 3 (Day 56).
  Interventions: Device: ELLIPTA placebo DPI; Device: DISKUS placebo DPI; Device: HandiHaler placebo DPI; Other: Inhaler preference questionnaires
- Treatment sequence C (Experimental): Eligible subjects will use DISKUS BID with HandiHaler QD for 28 days in Period 1 followed by ELLIPTA DPI QD use for 28 days in Period 2. These subjects will then be asked to complete preference questionnaire 1 at Visit 3 (Day 56).
  Interventions: Device: ELLIPTA placebo DPI; Device: DISKUS placebo DPI; Device: HandiHaler placebo DPI; Other: Inhaler preference questionnaires
- Treatment sequence D (Experimental): Eligible subjects will use DISKUS BID with HandiHaler QD for 28 days in Period 1 followed by ELLIPTA DPI QD use for 28 days in Period 2. These subjects will then be asked to complete preference questionnaire 2 at Visit 3 (Day 56).
  Interventions: Device: ELLIPTA placebo DPI; Device: DISKUS placebo DPI; Device: HandiHaler placebo DPI; Other: Inhaler preference questionnaires

INTERVENTIONS:
Device: ELLIPTA placebo DPI — ELLIPTA is a dry powder inhaler used via oral route. It will be a placebo DPI with two strips with 30 blisters per strip. First strip will contain lactose monohydrate and the second strip will contain lactose monohydrate blended with magnesium stearate.
Device: DISKUS placebo DPI — DISKUS is a dry powder inhaler used via oral route. It will be a placebo DPI with one blister strip that will contain lactose monohydrate.
Device: HandiHaler placebo DPI — HandiHaler is a dry powder inhaler used via oral route. It will be a DPI with placebo capsules that will contain lactose monohydrate.
Other: Inhaler preference questionnaires — Preference questionnaires will be given to subjects to understand the inhaler preference. There will be 2 types of questionnaire, preference questionnaires 1 and 2, which will be randomized at visit 3 (Day 56).

SUMMARY:
This randomized, cross over study aims to find out the benefits of delivering triple therapy using a single ELLIPTA® DPI (fixed-dose combination triple therapy) versus delivering triple therapy using two different types of inhalers (open triple therapy) including DISKUS® with HandiHaler® to subjects with COPD. Correct inhaler use, critical errors and performance attributes will also be assessed. Approximately 240 subjects with COPD will be randomized in the study. The study will be conducted in 3 visits and will be completed in approximately 56 days. At Visit 1 (Day 1) and Visit 2 (Day 28) subjects will be randomized to receive a placebo ELLIPTA inhaler once daily (QD) or a placebo DISKUS twice daily (BID) with placebo HandiHaler QD inhaler in 1:1 ratio in a cross-over manner for the study period (28 days for each period). At Visit 3 (Day 56), subjects will be asked to complete preference questionnaire 1 or 2. There will be no active treatment and subjects will continue to take their own prescribed COPD maintenance and rescue medication during the entire study period. ELLIPTA and DISKUS are the registered trademarks of GlaxoSmithKline group of companies. HandiHaler is the registered trademark of Boehringer Ingelheim group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be capable of giving signed informed consent.
* Subjects must have a diagnosis of COPD with a documented history of COPD for at least 12 months, in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Subjects must be 40 years of age inclusive, at the time of signing the informed consent.
* Male or female subjects will be included. Females must not be pregnant or planning pregnancy during the study or not lactating.
* Subjects must have a documented post albuterol forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) ratio <0.70 and FEV1 <=70% of predicted obtained within two years of Visit 1.
* Current or former (defined as subjects who have quit smoking for at least 3 months prior to Screening/Visit 1) cigarette smokers with a > 10 pack-year smoking history [Number of pack-years = (number of cigarettes per day/20) x number of years smoked (example, 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years].
* All subjects should be currently receiving maintenance treatment for COPD for at least 4 weeks prior to Randomization/Visit 1 and evaluated as unlikely to change COPD treatment within 4 weeks of Visit 1.
* All subjects should be able to stay on their prescribed maintenance COPD inhaler (s) without change throughout the entire treatment period.
* Subjects must be able to read, comprehend, and record information in English.

Exclusion Criteria:

* Subjects must not have a current diagnosis of asthma.
* Subjects must not have used the ELLIPTA, DISKUS, or HandiHaler inhalers in the 12 months prior to Visit 1.
* Subjects must not be receiving their current COPD medications with the ELLIPTA, DISKUS, or HandiHaler inhalers.
* Subjects must not be receiving only inhaled short-acting beta-adrenergic agonists, i.e., albuterol as their daily COPD therapy (as needed or regularly scheduled).
* Subjects must not have experienced more than 1 COPD exacerbation which required hospitalization in the 12 months prior to Visit 1.
* Subjects must not have a known or suspected history of alcohol or drug abuse within the last 2 years.
* Subjects must not have a history of hypersensitivity to any component of the study inhalers (example, lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Subjects with other respiratory disorders, including active tuberculosis, active lung cancer, sarcoidosis, lung fibrosis, pulmonary hypertension, or pulmonary disease (including but not confined to asthma, bronchiectasis with the need for treatment, cystic fibrosis, and bronchopulmonary dysplasia), interstitial lung diseases or other active pulmonary diseases.
* Subjects with historical, or current evidence of clinically significant or rapidly progressing or unstable cardiovascular, neurological, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or which would affect the analysis if the disease/condition exacerbated during the study will be excluded.
* Subjects with history of psychiatric disease, intellectual impairment, poor motivation or other conditions that will limit the validity of informed consent to participate in the study will be excluded.
* Subjects at risk of non-compliance, or unable to comply with the study procedures, or unable to continue their current medications.
* Subjects who have received an investigational drug and/or medical device/inhaler within 30 days of entry into this study (Screening/Visit 1), or within five drug half-lives of the investigational drug, whichever is longer.
* Subjects will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub investigator, study coordinator, or employee of the participating investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- United States (17):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Natchitoches, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Monroe, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20372

REFERENCES:
- [Background] Kerwin EM, Spangenthal S, Zvarich M, Millar V, Jain R, Collison K, Sharma R. ELLIPTA Versus DISKUS plus HandiHaler in COPD: A Randomized, Open-Label, Crossover Study in a Clinical Trial Setting. Chronic Obstr Pulm Dis. 2020 Apr;7(2):118-129. doi: 10.15326/jcopdf.7.2.2019.0153. PMID 32324983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, multi-center, open-label study comparing placebo ELLIPTA with placebo DISKUS + HandiHaler to assess correct inhaler use in participants with Chronic Obstructive Pulmonary Disease (COPD). A total of 17 centers across United States participated in the study.
Pre-assignment Details: Out of 240 randomized participants (par), 239 entered the study as 1 par was randomized in error. In order to minimize potential bias the order of placebo devices & order of responses, in preference questionnaire (PQ), was randomized in a crossover design. All par on study received placebo only & participant flow reflects this as the only treatment
Groups:
- ELLIPTA/DISKUS+HANDIHALER/Q1: Participants received placebo via ELLIPTA dry powder inhaler (DPI) in period 1 and DISKUS DPI + HandiHaler in period 2, followed by preference questionnaire (PQ) version 1. There was no active treatment and participants continued to take their own prescribed COPD medication and rescue medications for the duration of the study
- ELLIPTA/DISKUS+HANDIHALER/Q2: Participants received placebo via ELLIPTA DPI in period 1 and DISKUS DPI + HandiHaler in period 2, followed by PQ2. There was no active treatment and participants continued to take their own prescribed COPD medication and rescue medications for the duration of the study
- DISKUS+HANDIHALER/ELLIPTA/Q1: Participants received placebo via DISKUS DPI + HandiHaler in period 1 and ELLIPTA DPI in period 2, followed by PQ1. There was no active treatment and participants continued to take their own prescribed COPD medication and rescue medications for the duration of the study
- DISKUS+HANDIHALER/ELLIPTA/Q2: Participants received placebo via DISKUS DPI + HandiHaler in period 1 and ELLIPTA DPI in period 2, followed by PQ2. There was no active treatment and participants continued to take their own prescribed COPD medication and rescue medications for the duration of the study
Period: Period 1 (28 Days)
Arm/Group | ELLIPTA/DISKUS+HANDIHALER/Q1 | ELLIPTA/DISKUS+HANDIHALER/Q2 | DISKUS+HANDIHALER/ELLIPTA/Q1 | DISKUS+HANDIHALER/ELLIPTA/Q2
Started | 60 | 59 | 60 | 60
Completed | 58 | 57 | 59 | 58
Not Completed | 2 | 2 | 1 | 2
Not completed — Adverse Event | 1 | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Period: Period 2 (28 Days)
Arm/Group | ELLIPTA/DISKUS+HANDIHALER/Q1 | ELLIPTA/DISKUS+HANDIHALER/Q2 | DISKUS+HANDIHALER/ELLIPTA/Q1 | DISKUS+HANDIHALER/ELLIPTA/Q2
Started | 58 | 57 | 59 | 58
Completed | 57 | 56 | 57 | 55
Not Completed | 1 | 1 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants received placebo via ELLIPTA dry powder inhaler (DPI) or DISKUS DPI in combination with HandiHaler DPI based on the following treatment sequences: Treatment Sequence A (ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by PQ 1.); Treatment Sequence B (ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by PQ2); Treatment Sequence C (DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ1); or Treatment Sequence D (DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ2). Participants continued to take their own prescribed COPD medication and rescue medications for the entire 56-day study period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 131
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  African American/African Heritage | 23
  White - Arabic/North African Heritage | 3
  White - White/Caucasian/European Heritage | 213

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Zero Errors After 28 Days of Inhaler Use in Each Treatment Phase (Primary Estimand: Hypothetical)
Description: A checklist for correct use of each inhaler was developed in Patient Instruction Leaflets (PIL's). Participants were guided by trained health care provider (HCP) to demonstrate correct use of inhaler. Baseline assessment was conducted when participant initially dispensed the inhaler. Second assessment was conducted after each 28day dosing period. Correct Use Check list was completed by HCP at each visit. Primary hypothetical estimand is the estimate of treatment effect of all participants who stayed on their randomized study device sequence and did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. Participants could attend visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. Participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included
Time Frame: Up to Day 56
Population: Intent-to-treat (ITT) Population comprised of all randomized participants, excluding those who were randomized in error, and did not have at least one error assessment at Visit 1. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- ELLIPTA: Participants were randomized to use placebo via ELLIPTA in either period 1 or 2.
- DISKUS + HANDIHALER: Participants were randomized to use placebo via DISKUS + HANDIHALER in period 1 or 2.
Arm/Group | ELLIPTA | DISKUS + HANDIHALER
Number analyzed (Participants) | 217 | 217
Percentage of participants | 96 | 87
Statistical Analysis 1: Comparison: ELLIPTA vs DISKUS + HANDIHALER; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 6.88, 95% CI 2-sided [1.97 to 54.28] — Participants included in the model as fixed strata, treatment option was included in the exact statement and period included as fixed effects; There are three intercurrent events identified which could impact upon the estimand of interest: * The participant could withdraw from randomised study device sequence and therefore withdraw from the study * The participant could change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER; these subjects should have been withdrawn from the study according to the protocol. * The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. Rescue Medication use and change to maintenance COPD medication which is not delivered via ELLIPTA, DISKUS or HANDIHALER are not considered intercurrent events

2. Secondary Outcome: Number of Errors by Type for Each Inhaler After 28 Days of Use in Each Treatment Phase (Primary Estimand: Hypothetical)
Description: The occurrence of each type of error for each inhaler (ELLIPTA, DISKUS or HANDIHALER) were evaluated based on the information collected in Correct Use Checklists. Primary estimand is the treatment effect estimated in participants who stayed on their randomised study device sequence & did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. For primary estimand, a sensitivity analysis using Cochran-Mantel-Haenszel test was performed on participants with discordant results. Only those participants who completed error assessments for both randomized treatment groups & experienced no intercurrent events were included. The number of error is reported as NA for the type of error which was not applicable to the particular inhaler type
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Errors
Groups:
- DISKUS; HandiHaler: Participants were randomized to use placebo via DISKUS + HANDIHALER in period 1 or 2.
Arm/Group | ELLIPTA | DISKUS | HandiHaler
Number analyzed (Participants) | 217 | 217 | 217
Errors
  Par exhales while holding inhaler away from mouth | 6 | 9 | 14
  Par takes long steady deep breath in through mouth | 2 | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler
  Par breathes out slowly and gently | 1 | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler
  Par opened cover | NA — NA indicates error not applicable for that particular inhaler | 1 | NA — NA indicates error not applicable for that particular inhaler
  Par slid lever away from mouthpiece | NA — NA indicates error not applicable for that particular inhaler | 1 | NA — NA indicates error not applicable for that particular inhaler
  Par didn't tilt/shake device post dose preparation | NA — NA indicates error not applicable for that particular inhaler | 2 | 1
  Par took a quick deep breath through the Diskus | NA — NA indicates error not applicable for that particular inhaler | 1 | NA — NA indicates error not applicable for that particular inhaler
  Par removed Diskus from mouth,held breath for long | NA — NA indicates error not applicable for that particular inhaler | 2 | NA — NA indicates error not applicable for that particular inhaler
  Par breathed out slowly | NA — NA indicates error not applicable for that particular inhaler | 1 | NA — NA indicates error not applicable for that particular inhaler
  Par closed the cover of the inhaler | NA — NA indicates error not applicable for that particular inhaler | 2 | NA — NA indicates error not applicable for that particular inhaler
  Par did not exhale into the mouthpiece | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 10
  Par opened mouthpiece & center chamber is showing | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 1
  Par opened only 1 capsule from the blister card | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 5
  Par placed capsule in center chamber of inhaler | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 1
  Par pressed green piercing button&released button | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 4
  Par exhaled fully | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 7
  Par closed lips tightly around mouthpiece | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 9
  Par didn't block air intake vents with fingers | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 9
  Par breathed in deeply | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 10
  Par heard or felt the capsule vibrate | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 14
  Par held breath for few seconds & removed inhaler | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 10
  Par resumed normal breathing | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 9
  Par didn't pierce use capsule for 2nd inhalation | NA — NA indicates error not applicable for that particular inhaler | NA — NA indicates error not applicable for that particular inhaler | 1

3. Primary Outcome: Percentage of Participants With Atleast One Error After 28 Days of Inhaler Use in Each Treatment Phase (Primary Estimand: Hypothetical)
Description: Primary estimand is the treatment effect estimated in participants who stayed on their randomised study device sequence and did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. For primary estimand, a sensitivity analysis using Cochran-Mantel-Haenszel test was performed on participants with discordant results. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- All Study Participants: Participants received placebo via ELLIPTA dry powder inhaler (DPI) or DISKUS DPI in combination with HandiHaler DPI based on the following treatment sequences: Treatment Sequence A (ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by PQ 1.); Treatment Sequence B (ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by PQ2); Treatment Sequence C (DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ1); or Treatment Sequence D (DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ2). Participants continued to take their own prescribed COPD medication and rescue medications for the entire 56-day study period. All participants on study received placebo only and participant flow reflects this as the only treatment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 217
Percentage of participants
  Atleast 1 error-ELLIPTA&0 errors-DISKUS+HandiHaler | 3
  Atleast 1error-DISKUS+HandiHaler&0errors-ELLIPTA | 23
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Sensitivity Analyses (Primary Estimand: Hypothetical)

4. Secondary Outcome: Number of Errors Per Participant for Each Treatment Group After 28 Days of Use (Primary Estimand: Hypothetical)
Description: Participants were provided with PIL explaining correct use of inhaler. Overall error includes both critical and non-critical errors. Primary estimand is the treatment effect estimated in participants who stayed on their randomised study device sequence and did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. For primary estimand, a sensitivity analysis using Cochran-Mantel-Haenszel test was performed on participants with discordant results. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included.
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Median (Full Range); unit: Errors per participant
Arm/Group | ELLIPTA | DISKUS + HandiHaler
Number analyzed (Participants) | 217 | 217
Errors per participant | 0.0 [0 to 1] | 0.6 [0 to 9]

5. Secondary Outcome: Change in Errors Per Participant for Each Treatment Group After 28 Days of Use
Description: Assessment of errors was conducted by HCP trained in the correct inhaler use of the three inhalers based on the checklist of errors. The median number of overall errors made by per participant was assessed for ELLIPTA and DISKUS + HandiHaler both on Day 1 and Day 28 for each treatment group. The difference was calculated by subtracting values of Day 28 from Day1 for each treatment regimen. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included.
Time Frame: Day 1 and Day 28 of each treatment group
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Median (Full Range); unit: Errors per participant
Arm/Group | ELLIPTA | DISKUS + HandiHaler
Number analyzed (Participants) | 217 | 217
Errors per participant | 0.0 [-3 to 1] | 0.0 [-10 to 9]

6. Secondary Outcome: Number of Errors for Each Treatment Group in Participants With One or More Errors After 28 Days of Use (Primary Estimand: Hypothetical)
Description: Participants were provided with the PIL, explaining correct use of the inhaler. Overall error includes both critical and non-critical errors. Assessment of errors was conducted by HCP trained in the correct inhaler use of the three inhalers based on the checklist of errors. Primary estimand is the treatment effect estimated in participants who stayed on their randomised study device sequence and did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. For primary estimand, a sensitivity analysis using Cochran-Mantel-Haenszel test was performed on participants with discordant results. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included.
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Median (Full Range); unit: Errors per participant
Arm/Group | ELLIPTA | DISKUS + HandiHaler
Number analyzed (Participants) | 217 | 217
Errors per participant | 1.0 [1 to 1] | 4.4 [1 to 9]

7. Secondary Outcome: Change in Errors for Each Treatment Group in Participants With One or More Errors After 28 Days of Use
Description: Assessment of errors was conducted by health care professionals trained in the correct inhaler use of the three inhalers based on the checklist of errors. The median of overall errors made by each participant was assessed for ELLIPTA and DISKUS + HandiHaler both on Day 1 and Day 28. The difference was calculated by subtracting values of Day 28 from Day1 for each treatment regimen. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included.
Time Frame: Day 1 and Day 28 of each treatment group
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Median (Full Range); unit: Errors per participant
Arm/Group | ELLIPTA | DISKUS + HandiHaler
Number analyzed (Participants) | 217 | 217
Errors per participant | 0.7 [-1 to 1] | 2.6 [-4 to 9]

8. Secondary Outcome: Number of Participants With Zero Critical Errors After 28 Days of Each Treatment Group Use (Primary Estimand: Hypothetical)
Description: A checklist for correct use of each inhaler was developed based on the steps identified in the PIL. A critical error was defined as an error that was most likely to result in no, or a significantly reduced amount, of medication being inhaled by the participant. Primary estimand is the treatment effect estimated in participants who stayed on their randomised study device sequence and did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. For primary estimand, a sensitivity analysis using Cochran-Mantel-Haenszel test was performed on participants with discordant results. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included.
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | ELLIPTA | DISKUS + HandiHaler
Number analyzed (Participants) | 217 | 217
Participants | 215 | 193
Statistical Analysis 1: Comparison: ELLIPTA vs DISKUS + HandiHaler; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 8.85, 95% CI 2-sided [lower limit 3.45] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Percentage of Participants With Atleast One Error After 28 Days of Inhaler Use in Each Treatment Phase (Supplementary Estimand: Composite)
Description: Supplementary estimand estimated the composite effect of initial randomized treatment. A sensitivity analysis using the Cochran-Mantel-Haenszel test was performed on participants with discordant results. Participants who withdrew during period 2 were included in the analysis using early withdrawal data where available or imputation otherwise. Participants who experienced an intercurrent event in Period 1 were excluded from the analysis.
Time Frame: Up to Day 56
Measure: Number; unit: Percentage of participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 224
Percentage of participants
  Atleast 1 error-ELLIPTA&0 errors-DISKUS+HandiHaler | 4
  Atleast 1error-DISKUS+HandiHaler&0errors-ELLIPTA | 27
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Sensitivity Analyses (Supplementary Estimand: Composite)

10. Secondary Outcome: Number of Participants With Atleast One Critical Error After 28 Days of Each Treatment Group Use (Primary Estimand: Hypothetical)
Description: A critical error was defined as an error that was most likely to result in no, or a significantly reduced amount, of medication being inhaled by the participant. Primary estimand is the treatment effect estimated in participants who stayed on their randomised study device sequence and did not change their standard COPD maintenance medication device to one delivered via ELLIPTA, DISKUS or HANDIHALER, throughout both 28 day treatment periods. The participant could attend the visit without the device/s they were randomised to, in which case correct use cannot be assessed as described in the protocol. For primary estimand, a sensitivity analysis using Cochran-Mantel-Haenszel test was performed on participants with discordant results. Only those participants who completed error assessments for both randomized treatment groups and experienced no intercurrent events were included.
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 217
Participants
  Atleast 1 critical error with ELLIPTA | 1
  Atleast 1 critical error with DISKUS+HandiHaler | 23
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Sensitivity Analyses (Primary Estimand: Hypothetical)

11. Secondary Outcome: Number of Participants With Atleast One Critical Error After 28 Days of Each Treatment Group Use (Supplementary Estimand: Composite)
Description: as for outcome 9
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 217
Participants
  Atleast 1 error-ELLIPTA&0 errors-DISKUS+HandiHaler | 3
  Atleast 1error-DISKUS+HandiHaler&0errors-ELLIPTA | 27
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Sensitivity Analyses (Supplementary Composite Estimand)

12. Primary Outcome: Percentage of Participants With Zero Errors After 28 Days of Inhaler Use in Each Treatment Phase(Supplementary Estimand: Composite)
Description: Supplementary estimand estimated the composite effect of initial randomized treatment. The analysis was performed using stratified exact logistic model. Participants were included in the model as fixed strata, treatment option was included in the exact statement and period included as fixed effects. Participants who withdrew during period 2 were included in the analysis using early withdrawal data where available or imputation otherwise. Participants who experienced an intercurrent event in Period 1 were excluded from the analysis.
Time Frame: Up to Day 56
Population: ITT Population. Only those participants with data available at specified time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA | DISKUS + HandiHaler
Number analyzed (Participants) | 224 | 224
Percentage of participants | 95 | 85
Statistical Analysis 1: Comparison: ELLIPTA vs DISKUS + HandiHaler; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 6.06, 95% CI 2-sided [2.08 to 24.55] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Day 56
Description: Intent-to-Treat Population was used to collect Adverse Events. Since all participants received placebo as treatment, data has been clubbed for all the arms. The non-serious AEs are reported using a frequency threshold of >5%
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/239
Serious Adverse Events (participants affected / at risk) | 10/239
Other Adverse Events (participants affected / at risk) | 0/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=239)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03227445/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT03227445/SAP_001.pdf